CLINICAL TRIAL: NCT05730842
Title: A Phase 1, Open-label Study in Healthy Male Subjects of the Absorption, Metabolism, Excretion, and Pharmacokinetics of EDG-5506 and an Absolute Bioavailability Study Using Radiolabeled EDG-5506
Brief Title: Absorption, Metabolism, Excretion and Absolute Bioavailability of EDG-5506 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDG-5506-103
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteer; Muscular Dystrophies; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn
Keywords: Healthy Volunteer
MeSH Terms: conditions — Muscular Dystrophies; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A - AME (Experimental): Evaluation of absorption, metabolism, excretion and pharmacokinetics of a single oral dose of radiolabeled EDG-5506 in healthy male volunteers
  Interventions: Drug: Radiolabeled EDG-5506 Suspension
- Part B - aBA (Experimental): Evaluation of bioavailability of a single oral dose of EDG-5506 followed by a single intravenous dose of radiolabeled EDG-5506 in healthy male volunteers
  Interventions: Drug: EDG-5506 Tablet; Drug: Radiolabeled EDG-5506 Intravenous

INTERVENTIONS:
Drug: EDG-5506 Tablet — Single Oral Dose - Tablet
  Arms: Part B - aBA
Drug: Radiolabeled EDG-5506 Suspension — Single Oral Dose
  Arms: Part A - AME
Drug: Radiolabeled EDG-5506 Intravenous — Single Intravenous Dose
  Arms: Part B - aBA

SUMMARY:
This is a Phase 1 2-part, single-center, open-label study in healthy male volunteers. Part A will assess the absorption, metabolism, excretion, and pharmacokinetics of one oral dose of radiolabeled EDG-5506. Part B will assess bioavailability of EDG-5506 with a single oral dose of EDG-5506 and a single intravenous dose of radiolabeled EDG-5506.

DETAILED DESCRIPTION:
This is a Phase 1 2-part, single-center, open-label study.

Up to 15 (8 in Part A and 7 in Part B) healthy male subjects will be enrolled in the study.

Part A:

Potential subjects will be screened to assess eligibility within 28 days prior to dose administration. Subjects will be admitted on Day -1 and confined to the study site until at least Day 30. On Day 1, subjects will receive a single oral suspension. Blood, urine and feces samples will be collected for determination of EDG-5506 concentration, total radioactivity, and metabolite profiling and identification. Between Day 30 and Day 36, subjects will be discharged.

Part B:

Potential subjects will be screened to assess their eligibility within 42 days prior to dose administration. Subjects will be admitted on Day -1 and confined to the study site until Day 8. On Day 1, subjects will receive a single oral dose of EDG-5506 in the fasted state followed 2 hours later by a single dose of radiolabeled EDG-5506. Subjects will be discharged from the study site on Day 8. Blood samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. For both Part A and Part B, males, of any race, between 18 and 55 years of age, inclusive.
2. For both Part A and Part B, a body mass index between 18.0 and 32.0 kg/m2, inclusive, and a total body weight greater than or equal to 50 kg.
3. In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram, vital signs measurements, and clinical laboratory evaluations at screening and check-in.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, genitourinary, immunological, or psychiatric disorder, as determined by the investigator (or designee).
2. Participation in a clinical study involving administration of an investigational drug in the past 30 days or 5 half-lives (whichever is longer) prior to dosing.
3. Participation in more than 3 radiolabeled drug studies in the last 12 months.
4. Poor peripheral venous access.
5. Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial x-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
The mass balance of EDG-5506 as measured by the total radioactivity recovered in urine | Up to 37 days
The mass balance of EDG-5506 as measured by the total radioactivity recovered in feces | Up to 37 days
Plasma maximum measured drug concentration (Cmax) measurements for EDG-5506 | Up to 37 days
Characterization of EDG-5506 as measured by urinary recovery (fet1-t2) | Up to 37 days
Absolute bioavailability of EDG-5506 as measured by Fabs | Up to 9 days

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | Up to 37 days
Incidence of abnormal clinical laboratory test results | Up to 37 days
Incidence of abnormal electrocardiograms (ECGs) | Up to 37 days
Distribution of total radioactivity into blood cells as measured by whole blood to plasma concentration ratio | Up to 37 days

CONTACTS AND LOCATIONS:
Overall Officials: Sam Collins, MBBS, PhD, Study Chair — Edgewise Therapeutics, Inc.
Locations (1):
- Labcorp Clinical Research Unit, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No